CLINICAL TRIAL: NCT01041742
Title: Pulse Pressure Variation to Predict Fluid Responsiveness During Cardiac Displacement in Patients Undergoing Off-pump Coronary Artery Bypass Surgery
Brief Title: Pulse Pressure Variation (PPV) to Predict Fluid Responsiveness During Cardiac Displacement in Patients Undergoing Off-pump Coronary Artery Bypass Surgery (OPCAB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Yunseok Jeon, MD., Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-0910-047-297
Record Dates: First submitted 2009-12-30; First posted 2010-01-01 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPCAB (Experimental)
  Interventions: Procedure: fluid loading

INTERVENTIONS:
Procedure: fluid loading — fluid loading will be performed by using 6% hydroxyethyl starch solution , at 10 mL/kg.
  Other Names: HES 130/0.4; Voluven; Fresenius Kabe, Stans, Switzerland

SUMMARY:
Pulse pressure variation (PPV) known as a dynamic preload index is increasingly being used for guide of fluid management under various clinical situations. We hypothesized that PPV could play a role as a predictor of fluid responsiveness during displacement of the heart in patients undergoing off-pump coronary artery bypass surgery (OPCAB).

DETAILED DESCRIPTION:
The aim of this study was to investigate the ability of PPV to predict fluid responsiveness during displacement of the heart in patients undergoing off-pump coronary artery bypass surgery. After anesthesia, we will measure mean arterial pressure, heart rate, central venous pressure, mean pulmonary artery pressure, pulmonary arterial occlusion pressure, mixed venous oxygen saturation, PPV and cardiac index in patients receiving elective OPCAB. All parameters will be recorded at 5 minutes after the left anterior descending artery anastomosis, immediately after the displacement of the heart for the left circumflex artery anastomosis, and 10 minutes after fluid loading with hydroxyethyl starch 6%(10 mL/kg). Patients whose cardiac index increased by >15% to fluid loading will be defined as responders. To test the abilities of central venous pressure, pulmonary artery occlusion pressure and PPV to predict fluid responsiveness during heart displacement, areas under the receiver operating characteristics curves of the responders will be calculated and compared.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective off-pump coronary artery bypass surgery

Exclusion Criteria:

* unstable angina, preoperative arrhythmia, reduced ventricular function (ejection fraction < 40%), more than mild degree valvular heart disease, preoperative use of vasopressors or mechanical assist devices, intra-cardiac shunt, pulmonary artery hypertension, severe peripheral vascular obstructive disease, or esophageal pathology precluding the use of transesophageal echocardiography (TEE)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
pulse pressure variation | during displacement of the heart in OPCAB

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, MD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Jeon Y, Bahk JH, Gil NS, Kim KB, Hong DM, Kim HJ. Pulse-pressure variation predicts fluid responsiveness during heart displacement for off-pump coronary artery bypass surgery. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1056-62. doi: 10.1053/j.jvca.2011.07.013. Epub 2011 Sep 15. PMID 21924634